CLINICAL TRIAL: NCT00535561
Title: Iron Deficiency Anemia Can be an Indication for Treatment of Subclinical Hypothyroidism: A Randomized, Double Blinded Study
Brief Title: Iron Deficiency Anemia Can be an Indication for Treatment of Subclinical Hypothyroidism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duzce University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-5
Record Dates: First submitted 2007-09-25; First posted 2007-09-26 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Iron Deficiency Anemia; Subclinical Hypothyroidism
Keywords: iron deficiency anemia; anemia; hypothyroidism; subclinical hypothyroidism
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia; Hypothyroidism | interventions — ferrous sulfate; Thyroxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Oral iron treatment only- for iron deficiency anemia and subclinical hypothyroidism coexisting patients
  Interventions: Drug: Ferrous sulfate tablets 325 mg, po, TID
- 2 (Active Comparator): Oral iron plus levothyroxine treatment- for iron deficiency anemia and subclinical hypothyroidism coexisting patients
  Interventions: Drug: Ferrous sulfate plus levothyroxine

INTERVENTIONS:
Drug: Ferrous sulfate tablets 325 mg, po, TID
  Arms: 1
Drug: Ferrous sulfate plus levothyroxine — Combination of ferrous sulfate tablet 325mg plus levothyroxine tablet 25 micrograms, po, TID
  Arms: 2

SUMMARY:
To determine whether iron deficiency anemia can be an indication for the treatment of subclinical hypothyroidism.

DETAILED DESCRIPTION:
51 Patients presented to our university outpatient internal medicine clinic who are found to have iron deficiency anemia coexisting with subclinical hypothyroidism have been included in this study. Patients were randomly assigned to oral iron or oral iron plus levothyroxin therapy. The physician and the patients did not know who received oral iron only or oral iron plus levothyroxine treatment. Hematologic parameters as well as serum iron, ferritin and iron binding capacity were being measured at the beginning and 3 months after treatment in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis and laboratory confirmation of iron deficiency anemia and subclinical hypothyroidism
* Must be able to swallow tablets

Exclusion Criteria:

* Multifactorial anemia or anemia due to other reasons
* Iron deficiency anemia requiring urgent intervention- cardiac ischemia, severe anemia, GI or GU losses due to malignancy and or acute/subacute big loses by respiratory, Gİ, GU, etc. system
* Prior thyroid disorder and/or treatment history
* Presence of any other co-morbid disease like renal insufficiency/ failure, coronary heart disease, hypertension, diabetes mellitus, any endocrine system disease other than subclinical hypothyroidism

Ages: 23 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-06; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Significant improvement in Hgb and RBC | 3 months

SECONDARY OUTCOMES:
Significant improvement in serum iron, ferritin, TIBC and possibly in serum TSH and free T4 levels. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Cinemre, Assit. Prof., Study Director — Duzce University School of Medicine
Locations (1):
- Duzce University School of Medicine, Düzce, Turkey (Türkiye)

REFERENCES:
- [Background] Kong WM, Sheikh MH, Lumb PJ, Naoumova RP, Freedman DB, Crook M, Dore CJ, Finer N. A 6-month randomized trial of thyroxine treatment in women with mild subclinical hypothyroidism. Am J Med. 2002 Apr 1;112(5):348-54. doi: 10.1016/s0002-9343(02)01022-7. PMID 11904108
- [Background] Surks MI, Ortiz E, Daniels GH, Sawin CT, Col NF, Cobin RH, Franklyn JA, Hershman JM, Burman KD, Denke MA, Gorman C, Cooper RS, Weissman NJ. Subclinical thyroid disease: scientific review and guidelines for diagnosis and management. JAMA. 2004 Jan 14;291(2):228-38. doi: 10.1001/jama.291.2.228. PMID 14722150
- [Background] Horton L, Coburn RJ, England JM, Himsworth RL. The haematology of hypothyroidism. Q J Med. 1976 Jan;45(177):101-23. PMID 1257398
- [Background] Cooper DS. Clinical practice. Subclinical hypothyroidism. N Engl J Med. 2001 Jul 26;345(4):260-5. doi: 10.1056/NEJM200107263450406. No abstract available. PMID 11474665
- [Background] Gharib H, Tuttle RM, Baskin HJ, Fish LH, Singer PA, McDermott MT. Subclinical thyroid dysfunction: a joint statement on management from the American Association of Clinical Endocrinologists, the American Thyroid Association, and the Endocrine Society. J Clin Endocrinol Metab. 2005 Jan;90(1):581-5; discussion 586-7. doi: 10.1210/jc.2004-1231. No abstract available. PMID 15643019